CLINICAL TRIAL: NCT03042845
Title: Randomized Comparison of JUDkins vs tiGEr Catheter in Coronary Angiography Via the Right Radial Artery: the JUDGE Study
Acronym: JUDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Xanthopoulou Ioanna, Cardiologist, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUH1
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Judkins L3.5/R4 cardiac catheters (Active Comparator)
  Interventions: Device: Judkins 3.5L/4R cardiac catheters
- Tiger cardiac catheter (Experimental)
  Interventions: Device: Tiger cardiac catheter

INTERVENTIONS:
Device: Tiger cardiac catheter — Tiger cardiac catheter
  Arms: Tiger cardiac catheter
Device: Judkins 3.5L/4R cardiac catheters — Judkins 3.5L/4R cardiac catheters
  Arms: Judkins L3.5/R4 cardiac catheters

SUMMARY:
The investigators aim to assess safety and efficiency of Tiger II (5Fr; Terumo Interventional Systems, Somerset, New Jersey) vs Judkins (5Fr; 3.5L/4R, Medtronic Co) catheters, in coronary angiography via the right transradial route. This is a prospective, randomized, two-centre, study of parallel design. Consecutive patients with acute coronary syndrome (ACS), eligible for non-urgent coronary angiography, are randomized after successful cannulation of right radial artery and informed consent to either Tigger II or Judkins 3.5L/4R catheters.

DETAILED DESCRIPTION:
From the entrance of the first diagnostic catheter into the sheath and until the completion of the diagnostic coronary angiography will be the measurement of the endpoints of the study.

In case of failure to complete the coronary angiogram with the catheter study a crossover to the other catheter of the study will take place except in cases of severe spasm, where catheter choice will be at the discretion of the operator. In case of failure of the other study's catheter, next catheter's selection will be at operator's discretion. Patients included in the study, who do not process to adhoc PCI, will be monitored with baseline creatinine and creatinine value at day 2 or 3 after coronary angiography.

In all angiography films will be conducted offline analysis by two experienced operators for scoring opacification grade and coronary ostium contact with the catheters used.

DEFINITIONS Mild spasm Spasm causing well tolerated local pain Moderate spasm Spasm which causes severe pain but the handling of catheters remains satisfactory Severe spasm Spasm that leads to change diagnostic catheter or access site Duration of coronary angiogram Is defined as the time from the insertion of the first diagnostic coronary catheter in the sheath to the exit of the last diagnostic catheter from the sheath Radiation time Radiation time from the insertion of the first diagnostic coronary catheter in the right radial sheath to the exit of the last diagnostic catheter from the sheath Dose area product (DAP) DAP from the insertion of the first diagnostic coronary catheter in the sheath to the exit of the last diagnostic catheter from the sheath Contrast volume Contrast volume (ml) used from the insertion of the first diagnostic coronary catheter in the sheath to the exit of the last diagnostic catheter from the sheath Contrast induced nephropathy (CIN) Relative increase ≥25% from baseline or absolute increase ≥ 0.5mg/dl of serum creatinine within 48-72 hours of intravenous contrast administration Opacification grade 0=poor/non-diagnostic

1. moderate opacification only in systole or diastole
2. moderate opacification throughout cardiac cycle
3. complete opacification but not throughout cardiac cycle
4. complete opacification throughout cardiac cycle Catheter contact with coronary ostium

0=none and non-diagnostic study

1=none but diagnostic study 2=non-coaxial contact 3=coaxial contact Catheter stability within the coronary ostium 0=no catheter's steady engagement of the ostium throughout the angiographic view

1=catheter's steady engagement of the ostium throughout the angiographic view Catheter failure Completion of coronary angiogram after study catheter crossover with or without right radial access site crossover Based on pilot data and previously published data we hypothesized that Tiger catheter use will lead to an absolute decrease of at least 5 ml in contrast volume compared with Judkins catheters (48 and 53 ml for Tiger και Judkins catheters respectively, with estimated standard deviation of 17 for both). With a 2-sided alpha of 0.05, group sample sizes of 316 and 316 will achieve 95% power to detect this difference.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Indication for non-urgent coronary angiography
3. Successful cannulation of right radial artery
4. Availability of both Tiger and JL3.5/JR4 catheters

Exclusion Criteria

1. Indication for urgent coronary angiography (ST-elevation myocardial infarction or non ST-elevation myocardial infarction with indication for coronary angiogram within 2 hours)
2. Hemodynamic instability
3. Non palpable right coronary artery
4. Abnormal Allen test
5. Prior coronary artery bypass grafting
6. Chronic kidney disease or dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Contrast volume | End of coronary angiography
  Contrast volume (in ml) between groups used for completion of coronary angiogram in intention to treat analysis analysis

SECONDARY OUTCOMES:
Contrast volume | End of coronary angiography
  Contrast volume (in ml) between groups used for completion of coronary angiogram in per protocol analysis
Dose Area Product (DAP) | End of coronary angiography
  DAP (cGy*cm2) between groups in intention to treat and per protocol analysis
Fluoroscopy time | End of coronary angiography
  Fluoroscopy time (min) between groups in ITT and per protocol analysis
Contrast induced nephropathy (CIN) | End of coronary angiography
  CIN rate between groups in ITT and per protocol analysis
Catheter failure | End of coronary angiography
  Catheter failure rate between groups
Severe spasm | End of coronary angiography
  Severe spasm rate between groups
Coronary angiogram time | End of coronary angiography
  Duration of coronary angiogram between groups in ITT and per protocol analysis
Opacification grade | End of coronary angiography
  Opacification grade for LAD, LCX and RCA between study catheters
Contact to coronary ostium | End of coronary angiography
  Contact to left and right coronary ostium between study catheters
Stability within the coronary ostium | End of coronary angiography
  Catheter's steady engagement of the ostium throughout the angiographic view

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Patras University Hospital, Pátrai, Achaia
  - Second Department of Cardiology, Red Cross General Hospital, Athens

IPD SHARING:
Plan to Share IPD: Undecided